CLINICAL TRIAL: NCT00276224
Title: Iron Supplementation in Schistosomiasis and Soil Transmitted Helminths Control Programmes in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-ZM-VM-04
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Schistosomiasis; Helminthiases; Anaemia
Keywords: iron deficiency schistosomiasis soil transmitted helminths
MeSH Terms: conditions — Schistosomiasis; Helminthiasis; Anemia | interventions — ferrous sulfate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: ferrous sulphate (drug)

SUMMARY:
The objectives of this study is:

* to establish the coverage rate of weekly iron supplementation in children in intervention schools over a period of nine months
* document any side effects of weeekly iron supplementation among children in intervention schools over a period of nine months asses the feasibility of incorporating the weekly iron supplementation programme into the normal school activity in intervention schools determine the extent of acceptability and support for the iron supplementation programme by staff at the health centre nearest to the intervention schools
* compare the praziquantel efficacy and schistosomiasis reinfection in children in intervention schools with that of children in control schools following the introduction of weekely iron supplementation over a period of nine months
* determine the impact of weekly iron supplementation on haemoglobin levels of children in intervention schools and compare with children in control schools over a period of nine months

DETAILED DESCRIPTION:
Iron deficiency anaemia is a common denominator for both schistosomiasis and soil transmitted helminths. Iron deficiency appears to affect the immune response against schistosomes and intestinal helminths. It therefore follows that correcting the iron deficiency anaemia will improve the efficacy of anthelminthics such as praziquantel (against schistosomiasis) and albendazol (against soil transmitted helminths) and ability of the host immune system to resist reinfection with schistosomes and soil transmitted helminths.

The aim of this study is to identify factors necessary for a successful weekly iron supplementation programme in schistosomiasis and soil transmitted helminths control programmes. In addition impact of weekly iron supplementation programme n haemoglobin levels, efficacy of praziquantel, and schistosomiasis re-infection will be studied.

ELIGIBILITY:
Inclusion Criteria:all schoolchildren, in grade 2 and 3, at four selected schools -

Exclusion Criteria:

-

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480
Dates: Start 2005-09; Study Completion 2006-04

PRIMARY OUTCOMES:
Urine samples examined for schistsoma haematobium at month 0, 3. 6 and 9
Stool samples examined for schistsoma mansoni at mont 0, 3, 6 and 9
Blood samples examined for haemoglobin level mont 0 and month 9

SECONDARY OUTCOMES:
Any side effects to iron supplementation, measured every week for the first foru weeks after treatment start. Mesured on:
- headache
nausea
vomiting
body weakness
diarrhoea
abdominal pain
others

CONTACTS AND LOCATIONS:
Overall Officials: Victor Mwanakasale, Ph.d.,M.Sc., Principal Investigator — Tropical Disease Research Centre, Ndola, Zambia
Locations (1):
- Kenani and Chandwe School, Kenani, Nchelenge district, Zambia

REFERENCES:
- [Derived] Mwanakasale V, Siziya S, Mwansa J, Koukounari A, Fenwick A. Impact of iron supplementation on schistosomiasis control in Zambian school children in a highly endemic area. Malawi Med J. 2009 Mar;21(1):12-8. doi: 10.4314/mmj.v21i1.10982. PMID 19780472